CLINICAL TRIAL: NCT02733471
Title: Evaluation of the Efficacy and Safety of Administering Lidocaine Spray in Oesophago-gastro-duodenoscopy
Acronym: LIDOGTC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Irene Martin Marcos, Registered Nurse, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIDOGTC
Record Dates: First submitted 2016-03-02; First posted 2016-04-11 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Tolerance
Keywords: Lidocaine; Endoscopy; Tolerance
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Five lidocaine solution puffs (10mg lidocaine/puff) on the four posterior quadrants of the pharynx and on the base of the tongue, 3 minutes before the oesophago-gastro-duodenoscopy.
  Interventions: Drug: Lidocaine
- Control (Placebo Comparator): Five placebo solution puffs on the four posterior quadrants of the pharynx and on the base of the tongue, 3 minutes before the oesophago-gastro-duodenoscopy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
This study evaluates the efficacy and safety of the administration of lidocaine spray in oesophago-gastro-duodenoscopies. Half of the patients will receive lidocaine spray, while the other half will receive a placebo.

ELIGIBILITY:
Inclusion criteria:

* Patients aged over 18
* ASA I, II and III
* Non allergic to lidocaine or any of the drugs used in the study
* Consent form signed by the patient

Exclusion Criteria:

* Stomach or esophagus diagnosed cancer
* Giant hiatal hernia diagnosed
* Zenker's diverticulum diagnosed
* Achalasia diagnosed
* Patients aged over 70
* Medical history of moderate to severe liver disease
* Medical history of moderate to severe renal insufficiency
* Medical history of moderate to severe Obstructive Sleep Apnea Syndrome (OSA) (AHI≥15).
* Severe respiratory insufficiency(asmtha or COPD) diagnosed
* Patients with encephalopaty active
* Patients with medical history of methemoglobinemia
* Patients with history of drug abuse
* Patients with mental impairment
* Patients with BMI≥ 35
* Use of pediatric tube

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Degree of tolerance referred by the endoscopist in each group. | Up to 15 minutes after endoscopy
  Establish degree of tolerance referred by the endoscopist in each group according to the scale defined by Leich et al ( Gastrointestinal Endosc 1993;39:384-7)

SECONDARY OUTCOMES:
Degree of tolerance referred by the patient in each group | Up to 15 minutes after endoscopy
  Establish degree of tolerance referred by the patient in each group according to the scale defined by Leich et al
Endoscopist's level of satisfaction with the procedure in each group | Up to 15 minutes after endoscopy
  Endoscopist's level of satisfaction with the procedure according to a visual analogic scale
Patient's level of satisfaction with the procedure in each group. | Up to 15 minutes after endoscopy
  Patient's level of satisfaction with the procedure according to a visual analogic scale
Number of completed procedures in control and lidocaine group | Up to 15 minutes after endoscopy
  Number of completed procedures
Estimate the total dose of propofol used in each group | 15 minutes before endoscopy
  Dose of propofol used
Establish and compare the number of adverse events detected in control and lidocaine group | Up to 15 minutes after endoscopy
  Number of adverse events
Estimate the number of patients with retrograde amnesia in each group | Up to 15 minutes after endoscopy
  Number of patients referring retrograde amnesia
Estimate the number of patients with cough in each group | Up to 15 minutes after endoscopy
  Cough referred by the patient
Estimate the number of patients with oropharyngeal discomfort in each group. | Up to 15 minutes after endoscopy
  Oropharyngeal discomfort referred by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Irene Martin Marcos, RN, Principal Investigator — Basque Health System
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Alava, Spain

REFERENCES:
- [Derived] Martin-Marcos I, Fernandez-Morte N, Balsategui-Martin M, Ortiz-Cantero A, Bermudez-Ampudia C, Lopez-Picado A, Perez-Vaquero P, Salvador-Perez M, Cristobal-Dominguez E. Evaluation of pharyngeal lidocaine anesthesia for esophagogastroduodenoscopy: Double-blind randomized control trial. Dig Endosc. 2022 May;34(4):808-815. doi: 10.1111/den.14168. Epub 2021 Nov 17. PMID 34644419